CLINICAL TRIAL: NCT03802890
Title: Microbial Dysbiosis in the Pathogenesis of Rheumatoid Arthritis: Using Metagenomics to Predict Methotrexate Efficacy
Brief Title: Microbial Dysbiosis in Rheumatoid Arthritis
Acronym: MyRA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Action Arthritis (Other); University of East Anglia (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: QIB01/2018
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
Keywords: microbial dysbiosis; rheumatoid arthritis; dietary factors
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * faecal samples
  * blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MyRA study will primarily investigate whether there are associations between the structure and function of the gut microbiome and response to methotrexate in early rheumatoid arthritis patients. The microbiome will be characterised via shotgun metagenomic sequencing of microbial DNA present in stool samples taken during the participant's first 6 months of taking methotrexate.

DETAILED DESCRIPTION:
Methotrexate is often the first drug of choice for patients with early rheumatoid arthritis (RA), but its efficacy is highly variable and it can lead to severe side effects. There are currently no reliable predictors of methotrexate efficacy for people with early RA.

Microbial dysbiosis (an imbalanced microbiome) has recently been implicated in RA, with associations between specific microbes and RA biomarkers or disease activity. Gut microbes have extensive capabilities in terms of xenobiotic (e.g. drug) metabolism. Several gut microbes are able to alter the drug methotrexate in vitro, and it is possible this could effect drug efficacy in vivo. Alternatively methotrexate efficacy could be affected by baseline microbial composition or alterations to microbial composition over the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* RA diagnosis based on ACR 2010 classification criteria with symptoms starting within the last 2 years
* Referred by GP to the Early Arthritis Clinic at the Norfolk and Norwich University Hospitals NHS trust
* Commencing methotrexate monotherapy for the first time

Exclusion Criteria:

* Initially commencing combination therapy (prior to first stool sample) rather than methotrexate monotherapy i.e. MTX combined with another DMARD or prednisolone
* Commencement of MTX therapy prior to first stool sample or cessation of MTX therapy at any point during the study
* History of psoriasis
* Those currently suffering from, or have ever suffered from, any diagnosed gastrointestinal disease, gastrointestinal disorders including regular diarrhoea and constipation (excluding hiatus hernia unless symptomatic) and/or have undergone gastrointestinal surgery.
* Those regularly (3+ times/week) taking self-prescribed over the counter medications for digestive/gastrointestinal conditions
* Use of laxatives within 7 days prior to sampling unless these have been used on a regular basis (3+ times/week) for more than one month prior to the study and will continue to be used throughout the study period
* The use of over-the-counter medications or food/drinks containing pre and/or probiotics within 7 days prior to sampling, unless these have been used on a regular basis (3+ times/week) for more than one month prior to the study and will continue to be used throughout the study period
* Significant alteration of the participant's normal diet at any point during the study (e.g. adoption of the 5:2 fasting diet)
* Regular (3+ times/week) or recent (within 3 months) use of colonic irrigation or other bowel cleansing techniques
* Recently returned to the UK following a period abroad, and who have suffered gastric symptoms during the period abroad or on return to the UK. These will be assessed on an individual basis
* Currently taking or finished a course of antibiotics within the last 3 months
* Currently pregnant or lactating
* Living with or related to any member of the Study Team
* Those who have limited or no understanding of spoken and written English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early rheumatoid arthritis commencing methotrexate monotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in DAS28-CRP score | 0-6 months
  Disease Activity Score using 28 joints and C-reactive Protein

SECONDARY OUTCOMES:
Change in SDAI score | 0-6 months
  Simplified Disease Activity Index
Concentration of CRP in blood | 0-6 months
  C-reactive Protein (an inflammatory biomarker)
ESR value (blood) | 0-6 months
  Erythrocyte Sedimentation Rate (an inflammatory biomarker)
Concentration of anti-CCP in blood | 0-6 months
  Anti-Cyclic Citrullinated peptide (disease-specific antibody)
Concentration of RF in blood | 0-6 months
  Rheumatoid Factor (disease-specific antibody)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Carding, Prof, Study Chair — Quadram Institute Bioscience
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03802890/Prot_000.pdf